CLINICAL TRIAL: NCT04216433
Title: A Large Surgical Registry for Abdominal Aortic Aneurysms (AAA)
Acronym: AAA
Status: Completed | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 2012.00.591.A
Record Dates: First submitted 2019-08-12; First posted 2020-01-02 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-09

CONDITIONS: Abdominal Aortic Aneurism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: endovascular surgery — an innovative, less invasive procedure used to treat problems affecting the blood vessels, such as an aneurysm, which is a swelling or "ballooning" of the blood vessel. The surgery involves making a small incision near each hip to access the blood vessels.

SUMMARY:
In the spirit of improving patient safety and quality of healthcare in our region, the Dallas-Fort Worth Hospital Council Education and Research Foundation (Foundation) and Baylor Research Institute sought and obtained federal funding support (AHRQ grant) to develop an Abdominal Aortic Aneurism (AAA) surgery registry in North Texas. Participating centers will directly benefit from this project and will have access to a de-identified version of the registry data through their collaboration. These data may be used for quality improvement initiatives and/or to conduct your own research. In summary, this effort represents a substantial investment (with no costs to facilities) in improving outcomes for patients with AAA.

DETAILED DESCRIPTION:
Currently, little is known about who receives which type of surgery. What data are available are largely from single-centre studies, with study populations of a few hundred to a thousand patients, comparing outcomes for open and endovascular repair and collecting patient characteristic data largely for risk adjustment. Data on endovascular vs open AAA repair from the population-based registry will provide important information regarding the current use of these two treatment strategies, as well as allowing comparison of long-term outcomes for each according to different patient characteristics.

The proposed registry has the potential to provide means for internal quality assessment for the participating institutions. The de-identified registry will be made available to researchers at their request. This registry, focusing on AAA in the Dallas-Fort Worth metroplex, will provide data with the potential to improve treatments for more than 800,000 patients in the US.

ELIGIBILITY:
Inclusion Criteria:

* Men and women who received endovascular or open AAA repair (primary/secondary procedure codes: ICD-9=38.44 for open, ICD-9=39.71 for endovascular repair) at any of the 138 Dallas-Fort Worth area hospitals that report AAA data to the DFWHC Data Initiative.
* patients age 50 years old or older.

Exclusion Criteria:

* Patients with HIV and substance abuse
* Patients with substance abuse
* Patients > 50 years old

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women who received endovascular or open AAA repair (primary/secondary procedure codes: ICD-9=38.44 for open, ICD-9=39.71 for endovascular repair) at any of the 138 Dallas-Fort Worth area hospitals that report AAA data to the DFWHC Data Initiative.
Sampling Method: Non-Probability Sample
Enrollment: 394 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | 2000 to 2009
  time (in days) from first AAA surgery to death (any cause)
Time to re-operation | 2000 to 2009
  time (in days) from first AAA surgery to AAA re-operation
Time to rupture | 2000 to 2009
  time (in days) from first AAA surgery to AAA rupture

SECONDARY OUTCOMES:
Type of AAA surgery | day of surgery
  either open or endovascular AAA surgery

CONTACTS AND LOCATIONS:
Overall Officials: Robert Feldtman, MD, Principal Investigator — DFW Vascular Group
Locations (1):
- Methodist Health System, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided